CLINICAL TRIAL: NCT00140465
Title: A Double-Blind, Randomized Comparison Between Two Different Clopidogrel Maintenance Doses After Percutaneous Coronary Intervention (ISAR-CHOICE-2)
Brief Title: 75 or 150 mg Clopidogrel Maintenance Doses Following PCI (ISAR-CHOICE-2)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Technical University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GE IDE No. A00803
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 75 mg Clopidogrel Maintenance Doses
  Interventions: Drug: Clopidogrel
- 2 (Active Comparator): 150 mg Clopidogrel Maintenance Doses
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — after PCI
  Other Names: Iscover; Plavix
  Arms: 1
Drug: Clopidogrel — after PCI
  Other Names: Iscover; Plavix
  Arms: 2

SUMMARY:
The purpose of the study is to test whether an increase of the maintenance dose of clopidogrel from 75 to 150 mg per day results in an additional suppression of ADP-induced platelet aggregation

DETAILED DESCRIPTION:
In patients treated with coronary stents clopidogrel therapy is usually initiated with a 300 to 600 mg loading dose. In the CREDO trial it was shown that a 300 mg loading dose results in a reduction of ischemic events after percutaneous coronary intervention (PCI) if given 6 hours prior to the procedure. An antiplatelet effect similar to that achieved by chronic therapy with 75 mg/day is reached within 2 hours when the high 600 mg loading is administered. The 600 mg loading dose has been shown to be safe and effective in preventing thrombotic events following coronary stent implantation. Recently, it was shown that in patients with stable angina and administration of the 600 mg loading dose at least two hours prior to PCI concomitant therapy with a GP IIb/IIIa antagonist does not result in a further reduction of the incidence of thrombotic events. In contrast to a number of investigations with different loading doses, no trials have been performed comparing different clopidogrel maintenance doses. Recently, it was shown that administration of a 600 mg loading dose in patients already on chronic clopidogrel therapy (75 mg/day) results in an additional significant increase in inhibition of adenosine diphosphate (ADP-) induced platelet aggregation. Therefore, it is possible that an increase of the clopidogrel maintenance dose in patients with chronic clopidogrel therapy also results in a more pronounced inhibition of platelet aggregation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic aspirin therapy who are treated with percutaneous coronary intervention at least 2 hours after administration of a 600 mg loading dose of clopidogrel

Exclusion Criteria:

* Major alterations of blood count (particularly platelet count < 100x10^9/l, haemoglobin < 10 mg/dl
* Recent bleeding diathesis
* Presence of a hematologic or malignant disorder
* Oral anticoagulation with coumarin derivates
* Use of glycoprotein (GP) IIb/IIIa antagonists during the intervention or during the preceding 14 days
* Therapy with clopidogrel within the last 28 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-10; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Maximal ADP(5µmol/l)-induced platelet aggregation 30 days after the intervention | 30 days after the intervention

SECONDARY OUTCOMES:
Maximal ADP(20µmol/l)-induced platelet aggregation 30 days after the intervention | 30 days after the intervention
P2Y12 inhibition measured by point-of-care test | P2Y12 inhibition measured by point-of-care test

CONTACTS AND LOCATIONS:
Overall Officials: Albert Schomig, MD, Study Chair — Deutsches Herzzentrum Muenchen; Adnan Kastrati, MD, Study Director — Deutsches Herzzentrum Muenchen; Nicolas von Beckerath, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (1):
- Deutsches Herzzentrum Muenchen, Munich, Germany

REFERENCES:
- [Background] Steinhubl SR, Berger PB, Mann JT 3rd, Fry ET, DeLago A, Wilmer C, Topol EJ; CREDO Investigators. Clopidogrel for the Reduction of Events During Observation. Early and sustained dual oral antiplatelet therapy following percutaneous coronary intervention: a randomized controlled trial. JAMA. 2002 Nov 20;288(19):2411-20. doi: 10.1001/jama.288.19.2411. PMID 12435254
- [Background] Pache J, Kastrati A, Mehilli J, Gawaz M, Neumann FJ, Seyfarth M, Hall D, Braun S, Dirschinger J, Schomig A. Clopidogrel therapy in patients undergoing coronary stenting: value of a high-loading-dose regimen. Catheter Cardiovasc Interv. 2002 Apr;55(4):436-41. doi: 10.1002/ccd.10092. PMID 11948888
- [Background] Kastrati A, Mehilli J, Schuhlen H, Dirschinger J, Dotzer F, ten Berg JM, Neumann FJ, Bollwein H, Volmer C, Gawaz M, Berger PB, Schomig A; Intracoronary Stenting and Antithrombotic Regimen-Rapid Early Action for Coronary Treatment Study Investigators. A clinical trial of abciximab in elective percutaneous coronary intervention after pretreatment with clopidogrel. N Engl J Med. 2004 Jan 15;350(3):232-8. doi: 10.1056/NEJMoa031859. PMID 14724302
- [Background] Muller I, Seyfarth M, Rudiger S, Wolf B, Pogatsa-Murray G, Schomig A, Gawaz M. Effect of a high loading dose of clopidogrel on platelet function in patients undergoing coronary stent placement. Heart. 2001 Jan;85(1):92-3. doi: 10.1136/heart.85.1.92. No abstract available. PMID 11119474
- [Background] Braunwald E, Antman EM, Beasley JW, Califf RM, Cheitlin MD, Hochman JS, Jones RH, Kereiakes D, Kupersmith J, Levin TN, Pepine CJ, Schaeffer JW, Smith EE 3rd, Steward DE, Theroux P, Gibbons RJ, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Hiratzka LF, Jacobs AK, Smith SC Jr; American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee on the Management of Patients With Unstable Angina). ACC/AHA guideline update for the management of patients with unstable angina and non-ST-segment elevation myocardial infarction--2002: summary article: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee on the Management of Patients With Unstable Angina). Circulation. 2002 Oct 1;106(14):1893-900. doi: 10.1161/01.cir.0000037106.76139.53. No abstract available. PMID 12356647
- [Background] Gorchakova O, von Beckerath N, Gawaz M, Mocz A, Joost A, Schomig A, Kastrati A. Antiplatelet effects of a 600 mg loading dose of clopidogrel are not attenuated in patients receiving atorvastatin or simvastatin for at least 4 weeks prior to coronary artery stenting. Eur Heart J. 2004 Nov;25(21):1898-902. doi: 10.1016/j.ehj.2003.10.039. PMID 15522468
- [Background] Kastrati A, von Beckerath N, Joost A, Pogatsa-Murray G, Gorchakova O, Schomig A. Loading with 600 mg clopidogrel in patients with coronary artery disease with and without chronic clopidogrel therapy. Circulation. 2004 Oct 5;110(14):1916-9. doi: 10.1161/01.CIR.0000137972.74120.12. Epub 2004 Jul 19. PMID 15262828